CLINICAL TRIAL: NCT07088458
Title: An Observational Study to Learn More About How Well Damoctocog Alfa Pegol Works in Previously Treated Children With Hemophilia A
Acronym: HEM-POWR Kids
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22991
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Previously treated patients (PTPs) with hemophilia A: Previously treated patients with hemophilia A who have been prescribed damoctocog alfa pegol for regular continuous prophylaxis.
  Interventions: Drug: Damoctocog alfa pegol (Jivi, Bay94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, Bay94-9027) — Follow clinical practice of BAY94-9027 to further define the treatment outcomes of damoctocog alfa pegol based on real-world use for regular prophylaxis in ages 7 to <12 years, including a broader population and a real-world treatment patterns.

SUMMARY:
This is an observational study of children with mild, moderate, or severe hemophilia A who are receiving damoctocog alfa pegol, and are between 7 to <12 years of age at the time of enrolment. Observational studies use data that are collected as part of routine medical care and participants do not receive any advice or any changes to healthcare as part of the study.

In this study, the data will be collected from participants who are receiving their usual treatment with damoctocog alfa pegol as prescribed by their doctor. These children have previously received damoctocog alfa pegol or other factor 8 (FVIII) products.

Hemophilia A is a genetic bleeding disorder. It is caused by the lack of a protein called clotting factor 8 (FVIII) that helps blood to clot properly. Lack of FVIII can result in excessive blood loss or bleeding inside the body after being injured or having surgery. At times, there is spontaneous bleeding into the joint spaces that leads to joint damage.

The drug observed in this study, damoctocog alfa pegol, is approved for doctors to prescribe to children who are at least 7 years old with hemophilia A. It is used to prevent or treat bleeding episodes and works by replacing missing FVIII in the body of people with hemophilia A.

The participants will receive damoctocog alfa pegol as prescribed independently by their own doctors during routine practice, not as a part of the study. Participants may choose to enroll in the study at any time after their doctor has prescribed damoctocog alfa pegol to prevent bleeding episodes.

The main purpose of this study is to learn more about how a treatment with damoctocog alfa pegol works to prevent bleeding episodes in routine medical practice. To answer this question, doctors will collect:

* information about bleeding episodes including the type and the location of the bleed
* information about the treatment with damoctocog alfa pegol and other FVIII products
* the overall health status of the participants

Data will be collected from participants over two years after they enroll in the study or until they choose to leave the study or switch to another hemophilia A treatment. Historical data will come from the participants' medical records or by interviewing the patient and parent/ legal guardian. The children's parents/ guardians will be asked to maintain a health diary to record details of bleeding episodes and treatment with damoctocog alfa pegol. The children's parents/ guardians will also be asked to answer a questionnaire (Hemo QoL-SF and PedHAL) to assess the effect of hemophilia on their child's daily life.

In this study, only available data from routine care will be collected. No additional visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A
* Patients must be 7 to < 12 years of age at enrollment
* Patients previously treated for hemophilia A ((≥50 exposure days to FVIII)
* No current evidence of FVIII inhibitor or clinical suspicion of FVIII inhibitor
* Patients without a previous history of inhibitors or patients with a previous history of inhibitors on standard prophylaxis therapy for at least 1 year prior to study entry
* Initiation of prescription or currently prescribed damoctocog alfa pegol for regular continuous prophylaxis (intent to treat for 52 weeks/year)
* Signed informed consent/assent.

Exclusion Criteria:

* Presence of a FVIII inhibitor
* Concurrent participation in an investigational program with interventions outside of routine clinical practice
* Diagnosis of any other bleeding/coagulation disorder other than hemophilia A
* Use of another hemostatic agent as the primary method of bleeding prophylaxis during the observation period
* Contra-indications according to the local marketing authorization
* Current immune tolerance induction (ITI) treatment for a FVIII inhibitor

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients are to be enrolled from treatment centers specializing in the treatment of bleeding disorders in countries with market authorization for the use of damoctocog alfa pegol for patients aged >7 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of treated bleeds per individual diary documentation period while prescribed damoctocog alfa pegol prophylaxis (overall and by dosing regimen) | Up to 24 months

SECONDARY OUTCOMES:
Number of treated and all bleeds for the different bleed types (spontaneous, trauma, joint) per individual diary documentation period while prescribed damoctocog alfa pegol prophylaxis (overall and by dosing regimen) | Up to 24 months
Occurrence of bleeds during individual diary documentation period while prescribed damoctocog alfa pegol prophylaxis prescription (overall and by dosing regimen) | Up to 24 months
Occurrence of bleeds within 6 months' time intervals including the first and the last 6 months during observation period (overall and by dosing regimen) | Up to 24 months
Presence of target joints at enrollment and at end of prophylaxis prescription (overall and by dosing regimen) | Up to 24 months
Damoctocog alfa pegol dose per infusion (overall and by dosing regimen) | Up to 24 months
Number of FVIII infusions (overall and by dosing regimen) | Up to 24 months

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.